# **FULL TITLE OF THE STUDY**

Preoxygenation with high-flow nasal oxygen using Optiflow  $^{TM}$  - does speech have an effect on end-tidal oxygen achieved when compared to closed-mouth nasal breathing?

# SHORT STUDY TITLE

Preoxygenation with  $Optiflow^{TM}$  – the effect of speech on oxygenation.

### Statistical Analysis Plan

### Methods of randomisation

Participants were randomly allocated to the either the speech or non-speech arm of the study according to a random number generator and a key drawn up prior to randomisation. This was done following the consent and recruitment process to maintain allocation concealment. Figure 3. demonstrates the randomisation of participants.

| Number Generated | Assigned Group |
|------------------|----------------|
| Odd | Speech |
| Even | Non-speech |

Figure 3: A reference table to randomly allocate participants to both arms of the study.

#### **Power calculations**

The primary outcome measure was ETO<sub>2</sub> after 3 minutes of oxygen via the Optiflow<sup>TM</sup> device. In order to ascertain a sample size, data was taken from a previous study by J. Powell and P. Butler<sup>47</sup> showing that an ETO<sub>2</sub> of 0.85 could be achieved using the Optiflow device without speech. An estimate for the speech group was then decided (rendering an ETO<sub>2</sub> of 0.75, SD= 0.1) based off detecting a minimally significant difference. The sample size was generated by `G\*Power` software. This yielded a sample size of 28 whereby  $\alpha$ =0.05 and 1- $\beta$ =0.8. An unpaired t-test was performed, and all statistical analysis was carried out using GraphPad Prism 8.

### **Statistical Analysis**

The data was imported from an excel spreadsheet into GraphPad Prism 8. Prior to analysis, some normality tests were run to determine whether the data was parametric or non-parametric. 18 participants in the `Speech` group and 12 participants in the `Non-Speech` group were included in the analysis using parametric statistics for normally distributed data. The confidence intervals were set at 95% and a P value of <0.05 was used to confirm any statistical significance.

An unpaired t-test was then conducted to investigate the likelihood that the difference between the means had been caused by chance. This would help establish a relationship between  $ETO_2$  achieved at the end of three minutes between those in the speech arm compared against those in the non-speech arm.

To determine demographics, the mean (standard deviation) was used to calculate average age, whilst median and Interquartile range were used as a measure of distribution for BMI and height.